CLINICAL TRIAL: NCT05349812
Title: An Observational Study of Cxbladder Performance for Detection or Rule-out of Upper Tract Urothelial Cancer
Brief Title: Detection of Disease in the Upper Tract
Acronym: DEDUCT
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor focusing on completion of other studies at this time.
Sponsor: Pacific Edge Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: Pacificedgedx
Record Dates: First submitted 2022-04-18; First posted 2022-04-27 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2022-04

CONDITIONS: Upper Tract Urinary Carcinoma
Keywords: observational upper urinary tract carcinoma hematuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 30mls of freshly voided urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational study of Cxbladder performance for detection or rule-out of upper tract urothelial cancer. Subjects will be prospectively recruited to a single arm observational study to validate the performance characteristics of Cxbladder for suspected (UTUC) or for patients with a history of UTUC and are under surveillance for recurrence of disease.

DETAILED DESCRIPTION:
This is a single arm observational study prospectively recruiting eligible subjects with no apparent UC of the bladder following white light cystoscopy who have positive or suspicious urine cytology or imaging results.

Participants will undergo all clinical investigations as prescribed by the physician as per standard of care with addition of urine sampling to enable Cxbladder and central urine cytology testing. A mid-stream voided urine sample collected at the time of appointment will be used for Cxbladder and central urine cytology testing. Cxbladder and central cytology results will not be reported to the physician.

Urine sample testing will occur at Pacific Edge Ltd laboratories (Dunedin, New Zealand). Central urine cytology will be processed by an independent testing laboratory (Southern Community Laboratories, Dunedin, New Zealand). The remainder of the urine sample will be used for dipstick analysis of Specific Gravity, Leucocytes, Nitrites, Blood, Haemoglobin, and pH. The unused portion of this sample will be used for local cytology and any other analysis as deemed clinically appropriate. Central urine cytology results are not available to physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected to have UTUC following negative cystoscopy but positive or suspicious imaging and/or urine cytology.
2. Under surveillance for UTUC following a previous confirmed diagnosis of UTUC
3. Able to provide a voided urine sample of the required 30 ml minimum volume
4. Able to give written consent
5. Able and willing to comply with study requirement
6. Aged 18 years or older

Exclusion Criteria:

1. Prior genitourinary manipulation (flexible or rigid cystoscopy / catheterisation, urethral dilation) in the 14 days before urine collection
2. Total cystectomy of the bladder with bowel urinary diversion
3. Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a single arm observational study prospectively recruiting eligible patients with no apparent bladder cancer following white light cystoscopy but have positive or suspicious urine cytology or imaging results.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Performance of Cxbladder for the detection of Upper Tract Urothelial Carcinoma (UTUC) | Up to 36 months
  The number of subjects identified with UTUC by Cxbladder testing as verified by the gold standard for clinical diagnosis.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raman JD, Messer J, Sielatycki JA, Hollenbeak CS. Incidence and survival of patients with carcinoma of the ureter and renal pelvis in the USA, 1973-2005. BJU Int. 2011 Apr;107(7):1059-64. doi: 10.1111/j.1464-410X.2010.09675.x. Epub 2010 Sep 3. PMID 20825397
- [Background] Inman BA, Tran VT, Fradet Y, Lacombe L. Carcinoma of the upper urinary tract: predictors of survival and competing causes of mortality. Cancer. 2009 Jul 1;115(13):2853-62. doi: 10.1002/cncr.24339. PMID 19434668
- [Background] Cowan NC. CT urography for hematuria. Nat Rev Urol. 2012 Mar 13;9(4):218-26. doi: 10.1038/nrurol.2012.32. PMID 22410682
- [Background] Cowan NC, Turney BW, Taylor NJ, McCarthy CL, Crew JP. Multidetector computed tomography urography for diagnosing upper urinary tract urothelial tumour. BJU Int. 2007 Jun;99(6):1363-70. doi: 10.1111/j.1464-410X.2007.06766.x. Epub 2007 Apr 8. PMID 17428251
- [Background] Janisch F, Shariat SF, Baltzer P, Fajkovic H, Kimura S, Iwata T, Korn P, Yang L, Glybochko PV, Rink M, Abufaraj M. Diagnostic performance of multidetector computed tomographic (MDCTU) in upper tract urothelial carcinoma (UTUC): a systematic review and meta-analysis. World J Urol. 2020 May;38(5):1165-1175. doi: 10.1007/s00345-019-02875-8. Epub 2019 Jul 18. PMID 31321509
- [Background] Takahashi N, Glockner JF, Hartman RP, King BF, Leibovich BC, Stanley DW, Fitz-Gibbon PD, Kawashima A. Gadolinium enhanced magnetic resonance urography for upper urinary tract malignancy. J Urol. 2010 Apr;183(4):1330-65. doi: 10.1016/j.juro.2009.12.031. Epub 2010 Feb 19. PMID 20171676
- [Background] Freudenberg LS, Beyer T. Subjective perception of radiation risk. J Nucl Med. 2011 Dec;52 Suppl 2:29S-35S. doi: 10.2967/jnumed.110.085720. PMID 22144552
- [Background] Royal HD. Effects of low level radiation-what's new? Semin Nucl Med. 2008 Sep;38(5):392-402. doi: 10.1053/j.semnuclmed.2008.05.006. PMID 18662560
- [Background] Linet MS, Kim KP, Rajaraman P. Children's exposure to diagnostic medical radiation and cancer risk: epidemiologic and dosimetric considerations. Pediatr Radiol. 2009 Feb;39 Suppl 1(Suppl 1):S4-26. doi: 10.1007/s00247-008-1026-3. Epub 2008 Dec 16. PMID 19083224
- [Background] Mettler FA Jr, Huda W, Yoshizumi TT, Mahesh M. Effective doses in radiology and diagnostic nuclear medicine: a catalog. Radiology. 2008 Jul;248(1):254-63. doi: 10.1148/radiol.2481071451. PMID 18566177
- [Background] Amis ES Jr, Butler PF, Applegate KE, Birnbaum SB, Brateman LF, Hevezi JM, Mettler FA, Morin RL, Pentecost MJ, Smith GG, Strauss KJ, Zeman RK; American College of Radiology. American College of Radiology white paper on radiation dose in medicine. J Am Coll Radiol. 2007 May;4(5):272-84. doi: 10.1016/j.jacr.2007.03.002. PMID 17467608
- [Background] Messer J, Shariat SF, Brien JC, Herman MP, Ng CK, Scherr DS, Scoll B, Uzzo RG, Wille M, Eggener SE, Steinberg G, Terrell JD, Lucas SM, Lotan Y, Boorjian SA, Raman JD. Urinary cytology has a poor performance for predicting invasive or high-grade upper-tract urothelial carcinoma. BJU Int. 2011 Sep;108(5):701-5. doi: 10.1111/j.1464-410X.2010.09899.x. Epub 2011 Feb 14. PMID 21320275
- [Background] McHale T, Ohori NP, Cieply KM, Sherer C, Bastacky SI. Comparison of urinary cytology and fluorescence in situ hybridization in the detection of urothelial neoplasia: An analysis of discordant results. Diagn Cytopathol. 2019 Apr;47(4):282-288. doi: 10.1002/dc.24108. Epub 2018 Nov 12. PMID 30417563
- [Background] Johannes JR, Nelson E, Bibbo M, Bagley DH. Voided urine fluorescence in situ hybridization testing for upper tract urothelial carcinoma surveillance. J Urol. 2010 Sep;184(3):879-82. doi: 10.1016/j.juro.2010.05.023. PMID 20643443
- [Background] Kavalieris L, O'Sullivan PJ, Suttie JM, Pownall BK, Gilling PJ, Chemasle C, Darling DG. A segregation index combining phenotypic (clinical characteristics) and genotypic (gene expression) biomarkers from a urine sample to triage out patients presenting with hematuria who have a low probability of urothelial carcinoma. BMC Urol. 2015 Mar 27;15:23. doi: 10.1186/s12894-015-0018-5. PMID 25888331
- [Background] O'Sullivan P, Sharples K, Dalphin M, Davidson P, Gilling P, Cambridge L, Harvey J, Toro T, Giles N, Luxmanan C, Alves CF, Yoon HS, Hinder V, Masters J, Kennedy-Smith A, Beaven T, Guilford PJ. A multigene urine test for the detection and stratification of bladder cancer in patients presenting with hematuria. J Urol. 2012 Sep;188(3):741-7. doi: 10.1016/j.juro.2012.05.003. Epub 2012 Jul 19. PMID 22818138
- [Background] Kavalieris L, O'Sullivan P, Frampton C, Guilford P, Darling D, Jacobson E, Suttie J, Raman JD, Shariat SF, Lotan Y. Performance Characteristics of a Multigene Urine Biomarker Test for Monitoring for Recurrent Urothelial Carcinoma in a Multicenter Study. J Urol. 2017 Jun;197(6):1419-1426. doi: 10.1016/j.juro.2016.12.010. Epub 2016 Dec 14. PMID 27986532
- [Background] Lotan Y, O'Sullivan P, Raman JD, Shariat SF, Kavalieris L, Frampton C, Guilford P, Luxmanan C, Suttie J, Crist H, Scherr D, Asroff S, Goldfischer E, Thill J, Darling D. Clinical comparison of noninvasive urine tests for ruling out recurrent urothelial carcinoma. Urol Oncol. 2017 Aug;35(8):531.e15-531.e22. doi: 10.1016/j.urolonc.2017.03.008. Epub 2017 Mar 31. PMID 28366272
- [Background] Breen V, Kasabov N, Kamat AM, Jacobson E, Suttie JM, O'Sullivan PJ, Kavalieris L, Darling DG. A holistic comparative analysis of diagnostic tests for urothelial carcinoma: a study of Cxbladder Detect, UroVysion(R) FISH, NMP22(R) and cytology based on imputation of multiple datasets. BMC Med Res Methodol. 2015 May 12;15:45. doi: 10.1186/s12874-015-0036-8. PMID 25962444
- [Background] Mowatt G, Zhu S, Kilonzo M, Boachie C, Fraser C, Griffiths TR, N'Dow J, Nabi G, Cook J, Vale L. Systematic review of the clinical effectiveness and cost-effectiveness of photodynamic diagnosis and urine biomarkers (FISH, ImmunoCyt, NMP22) and cytology for the detection and follow-up of bladder cancer. Health Technol Assess. 2010 Jan;14(4):1-331, iii-iv. doi: 10.3310/hta14040. PMID 20082749
- [Background] Jocham D, Stepp H, Waidelich R. Photodynamic diagnosis in urology: state-of-the-art. Eur Urol. 2008 Jun;53(6):1138-48. doi: 10.1016/j.eururo.2007.11.048. Epub 2007 Dec 10. PMID 18096307
- [Background] Konety B, Shore N, Kader AK, Porten S, Daneshmand S, Lough T, Lotan Y. Evaluation of Cxbladder and Adjudication of Atypical Cytology and Equivocal Cystoscopy. Eur Urol. 2019 Aug;76(2):238-243. doi: 10.1016/j.eururo.2019.04.035. Epub 2019 May 16. PMID 31103391
- [Background] VandenBussche CJ, Allison DB, Gupta M, Ali SZ, Rosenthal DL. A 20-year and 46,000-specimen journey to Paris reveals the influence of reporting systems and passive peer feedback on pathologist practice patterns. Cancer Cytopathol. 2018 Jun;126(6):381-389. doi: 10.1002/cncy.22006. Epub 2018 May 14. PMID 29757495
- [Background] Koya M, Osborne S, Chemasle C, Porten S, Schuckman A, Kennedy-Smith A. An evaluation of the real world use and clinical utility of the Cxbladder Monitor assay in the follow-up of patients previously treated for bladder cancer. BMC Urol. 2020 Feb 11;20(1):12. doi: 10.1186/s12894-020-0583-0. PMID 32046687
- [Background] Davidson PJ, McGeoch G, Shand B. Assessment of a clinical pathway for investigation of haematuria that reduces the need for cystoscopy. N Z Med J. 2020 Dec 18;133(1527):71-82. PMID 33332329